CLINICAL TRIAL: NCT00738998
Title: Longitudinal Assessment of Arthralgia and Related Symptoms in Breast Cancer Patients Receiving Aromatase Inhibitors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Requested by PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-1038
Record Dates: First submitted 2008-08-13; First posted 2008-08-21 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Aromatase Inhibitors; Symptom Assessment; Questionnaire; Survey; Phone Call; Arimidex; Anastrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire and Telephone Assessments (Experimental): Breast cancer patients assigned to one or two groups: Group 1) enrolled at beginning of anastrozole treatment; or Group 2) if beginning third year of anastrozole treatment.
  Interventions: Behavioral: Questionnaire; Other: Phone Calls

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires about pain and other symptoms, quality of life, and ability to work will be completed.
  Other Names: Survey
Other: Phone Calls — A telephone system will call every 2 weeks so that you can rate your symptoms and how they interfere with daily activities. Each call will take about 5 minutes.

SUMMARY:
The goal of this research study is to learn more about what it is like for patients with breast cancer to receive treatment with the drug anastrozole. Researchers want to learn about possible symptoms, such as joint pain, that patients may experience during treatment. Researchers also want to learn more about which patients are most likely to have joint symptoms by looking at certain proteins from routine blood draw samples.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be assigned to one of two groups, depending on how long you have been receiving anastrozole treatment. If you are within two months prior to or one month after starting treatment, you will be assigned to Group 1 and you will be followed through 2 years of treatment. If you have been taking anastrozole for about 2 years, you will be assigned to Group 2 and you will be followed through your third year of treatment.

Study Procedures:

You will complete tests and procedures during your regularly scheduled clinic visits.

Assessment 1:

* You will be taught how to use an automated symptom assessment program. For this program, a telephone system will call you at your home at a time that is convenient for you. Using the numeric key pad on your telephone, you will rate your pain and how it interferes with your daily activities.
* You will complete questionnaires about your pain and other symptoms, quality of life, and your ability to work. Completing the questionnaires should take about 45 minutes.
* You will also complete some cognitive (mental) questionnaires that should take about 30 minutes to complete. The cognitive questionnaires will be given to learn about problems with attention or mental fatigue that may be related to your treatment. If you choose not to complete the cognitive questionnaires, you can still participate in this study.
* Blood (about 2 ½ tablespoons) will be drawn to learn about how certain proteins called cytokines (found in the blood) change during therapy. Researchers will also measure the C-reactive protein (CRP) which indicates whether there is inflammation in your body.
* You will have an exam of your bone joints and you will be shown how to perform a self-exam on your joints at home using a study joint pain kit. This kit will be mailed to you if you have a new joint pain.
* Demographic information (name, address, date of birth, weight, height, marital status, job status, education, medical insurance status, and race) will be collected.
* Participants in Group 2 will complete a medication adherence questionnaire. This questionnaire contains questions about the dose of anastrozole you are taking, if it has changed (increased or decreased), and if you have been given any drugs to help manage symptoms that you may be experiencing. This form should take about 5 minutes to complete.
* If your doctor in the breast clinic thinks you need to see a specialist because of the pain or swelling you are experiencing, you will be referred to a rheumatologist here at MD Anderson. The rheumatologist will perform a bone joint examination and may order a blood draw to test for inflammation in your body.

Telephone System Calls:

The telephone system will call you every 2 weeks at a time convenient to you so that you can rate your pain and how it interferes with your daily activities. Each phone call will take about 5 minutes to complete.

While you are on the study, if you report through the telephone system joint pain of a certain level of severity, a joint pain kit will be mailed to you along with a pre-addressed stamped envelope. Study staff will call you to let you know the kit is being mailed and that they can help you complete it, if needed. You will be asked to perform a self exam of your joints and to mark the area that is painful to you on the body drawing included in the kit. You will also answer some questions about your pain and about your medication and supplement use. You will be asked to return the completed kit to the project office in the pre-addressed stamped envelope included with the kit. This kit should be able to be completed in about 15 minutes.

Every Month:

The study coordinator will call you monthly at a time convenient to you so that you can rate your symptoms and how they interfere with your daily activities.

Every 4 - 6 Months:

Research staff will arrange to meet you at your regularly scheduled clinic visits. These visits will take about 45 minutes. At these visits, you will have the following exams:

* Demographic information (marital status, job status, education, weight, and medical insurance status will again be collected.
* Blood (about 2 ½ tablespoons) will be drawn for cytokines and CRP testing.
* You will be asked to complete some questionnaires about your symptoms, ability to work, and quality of life.
* All participants will repeat the medication adherence questionnaire.
* A brief exam of your bone joints will be performed by the research staff.
* You will be asked to tell researchers about any changes in the medications, both prescribed and over the counter, and supplements you may be taking.

Annual Visits:

At your regularly scheduled annual visit (up to 2 times while on study), you will complete the following tests:

-If you agreed at the beginning of the study, you will complete the cognitive questionnaires. This should take about 45 minutes to complete.

The entire study-related time you will spend at your annual visit will be about 1 hour and 30 minutes.

Research staff will also collect clinical information and test results from your medical record while you are on study.

Length of Study:

Participants in Group 1 will remain on the study for up to 2 years. Participants in Group 2 will remain on the study for 12-14 months, depending on how follow-up clinic visits are scheduled.

This is an investigational study. Up to 102 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with early stage hormone receptor positive breast cancer who are at these 2 time points in their anastrozole treatment: 1) at the time period between two months prior or one month after beginning of their anastrozole treatment (Cohort 1); 2) patients within +/- 2 months of the beginning of the third year of anastrozole treatment (Cohort 2).
2. Patients >= 18 years old.

Exclusion Criteria:

1. Patients with metastatic disease.
2. Patients who cannot complete the assessment tools.
3. Patients without telephone access.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2008-06-05 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence, onset and severity of arthralgia during anastrozole treatment | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cleeland, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org